CLINICAL TRIAL: NCT00208975
Title: Phase II Study of Fludarabine and Mitoxantrone, Followed by GM-CSF(Granulocyte-macrophage Colony-stimulating Factor) and Rituximab in Patients With Low Grade Non-Hodgkins Lymphoma: An Analysis of Efficacy and Tolerability
Brief Title: Phase II Study of Fludarabine and Mitoxantrone, Followed by GM-CSF(Granulocyte-macrophage Colony-stimulating Factor) and Rituximab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Emory University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Christopher R. Flowers, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1048-2001
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-05

CONDITIONS: Lymphoma
Keywords: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Mitoxantrone; Cyclophosphamide; fludarabine; Rituximab; Granulocyte-Macrophage Colony-Stimulating Factor; fludarabine phosphate; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fludarabine and Mitoxantrome followed by GM-CSF and Rituximab (Active Comparator): Initial patients (n=9) received fludarabine (25 mg/m2 IV) and mitoxantrone (10 mg/m2 IV)with sequential administration of GM-CSF (500 mcg subcutaneously) on days 6 and 7 and rituximab (375 mg/m2) on day 8.
  After a change in the protocol, all additional patients (n=6) received fludarabine (25 mg/m2 IV) and cyclophosphamide (250 mg/m2 IV)with sequential administration of GM-CSF (500 mcg subcutaneously) on days 6 and 7 and rituximab (375 mg/m2) on day 8. All patients received dditional doses of GM-CSF (days +8 through +14) were given for patients to reduce variability in neutropenic management.
  Interventions: Drug: Mitoxantrone/Cyclophosphamide, Fludarabine, Rituximab and GM-CSF

INTERVENTIONS:
Drug: Mitoxantrone/Cyclophosphamide, Fludarabine, Rituximab and GM-CSF — Initial patients (n=9) received fludarabine (25 mg/m^2 intravenously) and mitoxantrone (10 mg/m^2 intravenously)with sequential administration of GM-CSF(Granulocyte-macrophage colony stimulating factor) (500 µcg subcutaneously) on days 6 and 7 and rituximab (375 mg/m^2) on day 8.
  After a change in the protocol, all additional patients (n=6) received fludarabine (25 mg/m^2 intravenously) and cyclophosphamide (250 mg/m^2 intravenously)with sequential administration of GM-CSF (500 µcg subcutaneously) on days 6 and 7 and rituximab (375 mg/m^2) on day 8. All patients received additional doses of GM-CSF (days +8 through +14) were given for patients to reduce variability in neutropenic management.
  Other Names: Fludara, Sargramostim, Leukine, Rituxan

SUMMARY:
Patients with a low-grade, or indolent (slow-growing) form of non-Hodgkin's lymphoma (NHL) in which the usual survival is between 7-10 years are being asked to take part in this study. Although normally-used combinations of chemotherapy will cause NHL to disappear in 30-40% of patients (called complete response or complete remission), almost all will have their disease return.

In this study, researchers tested a combination of anti-cancer agents, fludarabine, rituximab and GM-CSF with mitoxantrone or cyclophosphamide to see if a better and more long-lasting response can be achieved. All of the medications are approved by the Food and Drug Administration (FDA) and are available on the market. The agents we will use are:

* Mitoxantrone and fludarabine and cyclophosphamide and fludarabine are combinations of chemotherapy drugs that have been successfully used to treat NHL/CLL (Chronic lymphocytic leukemia) that has returned after treatment and are comparable options for treatment.
* Rituximab, a monoclonal antibody that kills cancer cells by binding the CD20 antigen found on the surface of B-cells, commonly used along with chemotherapy drugs to improve response rates in lymphoma treatment.
* GM-CSF (granulocyte-macrophage colony stimulating factor, also called sargramostim, GM, or Leukine), a growth factor which stimulates the development of new ("stem") cells. GM-CSF encourages stem cells to divide, specialize, and become active. It is not a normal part of treatment for NHL.

Using GM-CSF in NHL treatment is the experimental part of this study. The main purpose of this study is to see if giving GM-CSF along with a standard anti-cancer treatment will work better to reduce cancer, and to look at side effects of the treatment.

DETAILED DESCRIPTION:
Patients with a low-grade, or indolent (slow-growing) form of non-Hodgkin's lymphoma (NHL) in which the usual survival is between 7-10 years are being asked to take part in this study. Although normally-used combinations of chemotherapy will cause NHL to disappear in 30-40% of patients (called complete response or complete remission), almost all will have their disease return.

When NHL is diagnosed, an abundance of white blood cells called B-lymphocytes (or B-cells) are found in the body. Almost all B-cells have a special protein on the surface called a CD20 antigen. Some anti-cancer drugs, called monoclonal antibodies, target cancer cells by binding, or "locking up", specific antigens found on their surfaces, which kills the cancer cells.

In this study, researchers will test a combination of anti-cancer agents to see if a better and more long-lasting response can be achieved. All of the medications are approved by the Food and Drug Administration (FDA) and are available on the market. The agents we will use are:

-Mitoxantrone and fludarabine, a combination of chemotherapy drugs that has been successfully used to treat NHL that has returned after treatment.

OR

* Cyclophosphamide and fludarabine, a combination of chemotherapy drugs that has been successfully used to treat NHL that has returned after treatment.
* Rituximab, a monoclonal antibody that kills cancer cells by binding the CD20 antigen found on the surface of B-cells, commonly used along with chemotherapy drugs to improve response rates in lymphoma treatment.
* GM-CSF (granulocyte-macrophage colony stimulating factor, also called sargramostim, GM, or Leukine), a growth factor which stimulates the development of new (stem) cells. GM-CSF encourages stem cells to divide, specialize, and become active. It is not a normal part of treatment for NHL.

Using GM-CSF in NHL treatment is the experimental part of this study. In studies done in the laboratory, GM-CSF caused an increase in the number of antigens, such as CD20, on the surface of B-cells. If more antigens are present, it may be easier to target cells that express CD20 or other antigens. Monoclonal antibodies (such as rituximab) might then be able to more effectively bind the antigens and kill the cancer cells.

The main purpose of this study is to see if giving GM-CSF along with a standard anti-cancer treatment will work better to reduce cancer, and to look at side effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* To qualify for this study, the patient must have relapsed, refractory or previously untreated low-grade (indolent) non-Hodgkin lymphoma of the following subtypes: Follicular center cell lymphoma grade 1, lymphoplasmacytoid lymphoma, small lymphocytic lymphoma, splenic marginal-zone types lymphoma, monocytoid B-cell lymphoma and extranodal mucosa-associated lymphoid tissue (MALT) lymphomas. Final eligibility will be determined by the health professionals conducting this clinical trial.

Exclusion Criteria:

* Patients who have received prior treatment with purine analogs will be excluded from this study. Also, patients whose diagnostic/histologic subtype cannot be confirmed by our institution will not be able to participate in this study. Final eligibility will be determined by the health professionals conducting this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-07; Primary Completion 2009-12 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Flowers, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Cohen JB, Bucur S, Winton EF, Sinha R, Heffner LT, King N, Lonial S, Langston AA, Waller EK, Hutchison-Rzepka A, Colbert A, Lechowicz MJ, Flowers CR. Combination of GM-CSF With Fludarabine-Containing Regimens in Chronic Lymphocytic Leukemia and Indolent Non-Hodgkin Lymphoma. Clin Lymphoma Myeloma Leuk. 2015 Sep;15(9):514-8. doi: 10.1016/j.clml.2015.06.009. Epub 2015 Jul 3. PMID 26297176

RESULTS

PARTICIPANT FLOW:
Groups:
- Fludarabine and Cyclophosphamide With Sequential Administratio: Patients will receive fludarabine and cyclophosphamide with sequential administration of GM-CSF on days 6 and 7 and rituximab on day 8.
Period: Overall Study
Arm/Group | Fludarabine and Cyclophosphamide With Sequential Administratio
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fludarabine and Cyclophosphamide With Sequential Administratio
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 6
Age Continuous [Median (Full Range); unit: years] | 62 [45 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 15
Diagnosis Type [Number; unit: Participants]
  Low Grade Non Hodgkin's Lymphoma(NHL) | 7
  Chronic Lymphocytic Leukemia (CLL) | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients's Who Had Complete Response and Partial Response to the Treatment of Fludarabine and Cyclophosphamide Followed by GM-CSF and Rituximab.
Description: Complete Response (CR): Disappearance of all clinical evidence of active tumor for a minimum of eight weeks and absence of any symptoms related to the tumor.
  Partial Response (PR):50% decrease in the sum of the product diameters of all lesions that persist for at least four weeks. No lesion can increase in size and no new lesion can appear during this period.
  Stable disease (SD):A tumor that is neither growing nor shrinking.No new tumors have developed
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Chronic Lymphocytic Leukemia: Chronic Lymphocytic Leukemia (CLL) is a condition characterized by an accumulation of abnormal lymphocytes in the blood and the bone marrow. These lymphocytes do not perform their functions as normal ones would and interfere with the production of other blood cells necessary for the normal functioning of the blood, leading to a host of complications like deficiency of the immune system, coagulation problems, swollen lymph nodes, and many other conditions.
  Fludarabine-based combination provide effective treatment for patients with low-grade NHL and CLL with high complete response rates that are improved with the addition of Rituximab.
- Non Hodgkin Lymphoma: Non-Hodgkin's lymphoma, also called non-Hodgkin lymphoma, is cancer that originates in your lymphatic system, the disease-fighting network spread throughout your body. In non-Hodgkin's lymphoma, tumors develop from lymphocytes - a type of white blood cell.
  Fludarabine-based combination provide effective treatment for patients with low-grade NHL and CLL with high complete response rates that are improved with the addition of Rituximab.
Arm/Group | Chronic Lymphocytic Leukemia | Non Hodgkin Lymphoma
Number analyzed (Participants) | 8 | 7
participants
  Complete Response | 4 | 5
  Partial Response | 2 | 2
  Stable Disease | 1 | 0

ADVERSE EVENTS:
Arm/Group | Fludarabine and Cyclophosphamide With Sequential Administratio
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine and Cyclophosphamide With Sequential Administratio (N=15)
Neutropenia (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Anemia (Blood and lymphatic system disorders) | 9
Nausea (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 7
Vomiting (Gastrointestinal disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Fever (General disorders) | 3
Night Sweats (General disorders) | 4
Hyperkalemia (Renal and urinary disorders) | 1
Pain (General disorders) | 12
Constipation (Gastrointestinal disorders) | 5
Infusion reaction (Skin and subcutaneous tissue disorders) | 4
Hypoprotinemia (Blood and lymphatic system disorders) | 1
Weight Loss (General disorders) | 2
Loss of Appetite (General disorders) | 4
Anxiety (General disorders) | 2
Muscositis (Gastrointestinal disorders) | 3
Polyuria (Renal and urinary disorders) | 2
Hyperglycemia (Endocrine disorders) | 4
Malaise (General disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2

LIMITATIONS AND CAVEATS:
The protocol was closed early due to slow and poor accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes